CLINICAL TRIAL: NCT06040814
Title: To Explore the Changes of Fecal Microbiota Before and After Treatment in Patients With Liver Cirrhosis Complicated With Hepatic Encephalopathy or Sarcopenia as a Reference for Future Fecal Microbiota Transplantation
Brief Title: Microbiota, Sarcopenia, and Hepatic Encephalopathy Change in Cirrhotic Patients Before and After Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202201561B0
Record Dates: First submitted 2023-08-08; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2022-12

CONDITIONS: Hepatic Encephalopathy
Keywords: Liver cirrhosis; Hepatic encephalopathy; Psychometric test; Sarcopenia; Fecal microbiota
MeSH Terms: conditions — Hepatic Encephalopathy; Liver Cirrhosis; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation Training (Experimental): Rehabilitation Training is provided to patients with Liver Cirrhosis combined with sarcopenia.
  Interventions: Behavioral: Rehabilitation Training
- No-Rehabilitation Training (No Intervention): No extra training is provided to patients with Liver Cirrhosis combined with sarcopenia.

INTERVENTIONS:
Behavioral: Rehabilitation Training — 12 week Rehabilitation Training course
  Arms: Rehabilitation Training

SUMMARY:
Through this plan, it will provide many benefits to patients with liver cirrhosis complicated with sarcopenia and/or hepatic encephalopathy, their family members, and the government in Taiwan:

1. To explore the changes of fecal microbiota before and after treatment such as resistance training rehabilitation in patients with liver cirrhosis complicated with sarcopenia and/or hepatic encephalopathy as a reference for future fecal microbiota transplantation;
2. To measure the changes of sarcopenia level before and after rehabilitation;
3. To measure the changes of hepatic encephalopathy level before and after rehabilitation.

These study results will certainly bring updated diagnostic tool, latest treatment options, avoid serious sequelae and reduce medical expenditure.

DETAILED DESCRIPTION:
Chronic liver disease is notorious as Taiwan's national disease and more than 4,000 patients died of liver cirrhosis each year in Taiwan. Hepatic encephalopathy (HE) manifests from minimal HE (MHE) to overt HE (OHE). The diagnosis of covert HE (CHE) requires psychometric tests or neurophysiological tools. However, psychometric testing for patients with CHE is often neglected in Taiwan. On the basis of the capability to detect all forms of HE, further investigation on the association of HE with fecal microbiota alterations is urgently needed. It is because HE is associated with dysregulation in the gut-liver-brain axis, which includes intestinal barrier dysfunction and gut microbial dysbiosis. However, despite current standard of care (SOC) therapy i.e., lactulose and rifaximin, there remains a subset of patients who continue to suffer recurrence, which leads to further cognitive impairment, sarcopenia and readmissions. There remain several factors that can influence the microbiota, such as demographics (geographic area, sex and diet), etiology, drugs, interventions, and ﬁnally the sampling compartment. These factors need to be controlled for and considered in the interpretation of future studies. The microbiome dynamic change during rehabilitation in cirrhotic patients with sarcopenia has never been studied and is worth exploring.

Furthermore, from our previous study, the investigators have shown that one-year efficacy of rifaximin add-on to lactulose is superior to lactulose alone in patients with cirrhosis complicated with recurrent HE in Taiwan. The investigators also have preliminary data showing that rehabilitation could improve patient's sarcopenia. Further cohort validation is urgently required.

Our innovative research purposes:

1. To explore the changes of fecal microbiota before and after treatment such as resistance training rehabilitation as a reference for future fecal microbiota transplantation;
2. To measure the changes of sarcopenia levels before and after rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver cirrhosis

Exclusion Criteria:

* unstable vital sign such as shock, coma or intubation status
* Non-curative hepatocellular carcinoma (cannot receive operation, radiofrequency ablation, liver transplantation,etc
* Un-curative malignancies
* Poor-controlled diabetes mellitus (HbA1C≧8)
* Active alcoholism (male alcohol ≧40g/day, or ≧140g/week; female ≧ 30g/day, or ≧70g/week
* Psychiatric comorbidities
* Neurologic comorbidities like Alzheimer's, Parkinson's, stroke with neurological deficit
* Unable to speak
* Bed-ridden status
* Post- Liver transplantation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Handgrip Strength | 6 months
  Handgrip strength is an assessment of muscle strength. The cutoff value of the handgrip is < 30 kg in men and < 20 kg in women.
Short Physical Performance Battery (SPPB) | 6 months
  Short Physical Performance Battery (SPPB) is an assessment of physical performance. The cut-off value of the Short Physical Performance Battery (SPPB) score for determining sarcopenia is ≤ 9.
Dual-energy X-ray absorptiometry (DEXA) | 6 months
  Dual-energy X-ray absorptiometry (DXA) is the gold-standard technique in the analysis of body composition. The cut-off value of appendicular skeletal muscle mass (ASMI) score for determining sarcopenia is < 7.0 kg/m^2 in men and < 5.4 kg/m^2 in women.
Mini-Mental Status Examination (MMSE) | 6 months
  Mini-Mental State Examination (MMSE) is one of the most commonly used methods in the assessment of cognitive mental status. The cut-off value of Mini-Mental State Examination (MMSE) score is < 28.
Psychometric Hepatic Encephalopathy Score (PHES) | 6 months
  The psychometric hepatic encephalopathy score (PHES) is the gold standard for diagnosing minimal hepatic encephalopathy (MHE). The cut-off value of the Psychometric Hepatic Encephalopathy Score (PHES) for determining minimal hepatic encephalopathy (MHE) is ≤ -4.
Animal Naming Test (ANT) | 6 months
  The animal naming test (ANT) is an easy tool for the assessment of hepatic encephalopathy (HE). The cut-off value of the Animal Naming Test (ANT) score for determining hepatic encephalopathy (HE) is ≤ 19.
Blood cytokine levels [IL-6] | 6 months
  Serum IL-6 level (pg/ mL)
Blood ammonia levels [NH3] | 6 months
  Serum ammonia level (μg/dL)
Electroencephalogram (EEG) | 6 months
  Quantified EEG spectral analysis:
  Grade 0: Mean dominant frequency (MDF)> 6.8 Hz and no theta nor delta wave Grade 1: MDF > 6.8Hz and theta wave relative power ≧35% Grade 2: MDF≤ 6.8 Hz and delta wave relative power<49% Grade 3: MDF≤ 6.8 Hz and delta wave relative power≧49%
Fecal Microbiota | 6 months
  Check fecal microbiota taxonomy profile and relative abundance changes.

CONTACTS AND LOCATIONS:
Overall Officials: CHIEN-HAO HUANG, Principal Investigator — Linkou Chang Gung Memorial Hospital, Taoyuan, Taiwan
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No